

#### **Informed Consent**

Medical Record Number

INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Study of F18 Fluciclovine PET CT for Assessment of High-grade Glioma Tumor Volume and Radiation Response 2018-0869

Study Chair: Jason Johnson

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is

#### STUDY SUMMARY

provided after the summary.

Participant's Name

The goal of this clinical research study is to learn if a radioactive imaging agent called F18 Fluciclovine used during a PET-CT scan can help measure tumor size compared to standard of care MRI contrast agents, T2 FLAIR and T1, in patients with high-grade glioma who are having surgery to remove the tumor and are receiving radiation therapy.

F18 Fluciclovine is FDA-approved and commercially available radioactive imaging agent for PET scan in adult males with suspected prostate cancer. The PET-CT and MRI scans are performed using FDA approved and commercially available methods. Its use in this study is investigational.

Future patients may benefit from what is learned. There are no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

You can read a full list of potential side effects below in the Possible Risks section of this consent.

Your active participation in this study will be over after the 6-month scan.

The F18 Fluciclovine PET-CT and standard of care MRI scans will be performed at no cost to you while taking part in this study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive standard treatment for the disease. You may choose not to take part in this study. In all cases, you will receive appropriate medical care, including treatment for pain and symptoms of cancer.

#### 1. STUDY DETAILS

If you agree to take part in this study you will have 4 F18 Fluciclovine PET-CT scans paired with 4 standard of care MRI examinations (8 imaging scans total).

Up to 25 participants will be enrolled in this study. All will take part at MD Anderson.

You will have a F18 Fluciclovine PET-CT scan at the below time points. You will receive an injection of F18 Fluciclovine into a vein through a standard catheter while you lie in the scanner. The total PET-CT scan time is about 10 minutes.

- Within 14 days before the first standard of care tumor removal.
- Within 14 days before starting radiation therapy.
- About 21-35 days after finishing radiation therapy.
- About  $5\frac{1}{2}$   $6\frac{1}{2}$  months after finishing radiation therapy.

Within 3 days of each F18 Fluciclovine PET-CT scan, you will have a standard of care MRI of the brain with and without contrast. The total MRI scan time is about 45 minutes.

Your active participation in this study will be over after the 6-month F18 PET-CT scan. If you have follow-up MRIs as part of your standard care, about 3 and 6 months after your last study visit, the results of those MRIs will be collected.

### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The known side effects are listed in this form, but they will vary from person to person.

A **PET-CT scan** may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort or the scanning will be stopped.

The PET-CT scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing

them to radiation. You should drink fluids after the scan to help remove the solution from your system.

**18F Fluciclovine** may cause a feeling of warmth or pain at the injection site. They may cause nausea, vomiting, headache, dizziness, and/or heart and kidney complications. They may cause hypersensitivity reactions which may cause breathing and/or skin problems (rash, redness, blisters, itching, and/or local swellings) and may appear either immediately or up to a few days after the injection. It may cause water to collect in the lungs and/or anaphylactic shock (a severe allergic reaction that can cause breathing difficulty and/or a drop in blood pressure). It may cause changes in the way you move or changes in your senses.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

This study may involve unpredictable risks to the participants.

### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-2933 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the

research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

# **Additional Information**

- 4. You may ask the study chair (Dr. Jason Johnson, at 713-792-8443) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-2933 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor. If you withdraw from this study, you can still choose to be treated at MD Anderson.
- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study, including the results of all of your standard tests performed as part of this research, and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
  - The results of your imaging studies will be available to you after review by your primary physician.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.

### **Future Research**

Your personal information is being collected as part of this study. This information, or data, may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

Before being shared for future research, every effort will be made to remove your identifying information from any data. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data.

# **Authorization for Use and Disclosure of Protected Health Information (PHI):**

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form
- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.

E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think

about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT LEGALLY AUTHORIZED REPRESENTATIVE (LAR) The following signature line should only be filled out when the participant does not have the capacity to legally consent to take part in the study and/or sign this document on his or her own behalf. SIGNATURE OF LAR DATE PRINTED NAME and RELATIONSHIP TO PARTICIPANT WITNESS TO CONSENT I was present during the explanation of the research to be performed under Protocol 2018-0869. SIGNATURE OF WITNESS TO THE VERBAL CONSENT DATE PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for vulnerable adult participants. If witnessing the assent of a pediatric participant, leave this line blank and sign on the witness to assent page instead. PRINTED NAME OF WITNESS TO THE VERBAL CONSENT PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or her authorized representative, using language that is understandable and appropriate. I believe that I have fully informed this participant of the nature of this study and its possible benefits and risks and that the participant understood this explanation. PERSON OBTAINING CONSENT DATE PRINTED NAME OF PERSON OBTAINING CONSENT

# **TRANSLATOR**

| subtractions) into | nsent as written (without ad<br>and assisted | |
|---|---|---|
| (Name of Lange | | |
| obtaining and providing consent by tran | islating all questions and res | sponses during the consent |
| process for this participant. | | |
| | | <u> </u> |
| NAME OF TRANSLATOR SIGNAT | URE OF TRANSLATOR | DATE |
| ☐ Please check here if the translator witness, other than the translator, must | | • |
| SIGNATURE OF WITNESS TO THE V<br>(OTHER THAN TRANSLATOR, PAREI<br>OR STUDY CHAIR) | | DATE |
| ON OTODI OTIAIN) | | |
| PRINTED NAME OF WITNESS TO TH | E VERBAL TRANSLATION | |